CLINICAL TRIAL: NCT02904226
Title: Phase 1/2 Multicenter Trial of ICOS Agonist Monoclonal Antibody (mAb) JTX-2011 Alone and in Combination With Nivolumab, Ipilimumab, or Pembrolizumab in Adult Subjects With Advanced and/or Refractory Solid Tumor Malignancies
Brief Title: JTX-2011 Alone and in Combination With Anti-PD-1 or Anti-CTLA-4 in Subjects With Advanced and/or Refractory Solid Tumors
Acronym: ICONIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JTX-2011-101
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: ICOS; ICOS agonist monoclonal antibody; JTX-2011; Anti-PD-1; Nivolumab; ICONIC; Immunotherapy; Immuno-oncology; Cancer; Solid Tumor; Dose Escalation; Dose Expansion; Anti-CTLA-4; Ipilimumab; Pembrolizumab
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; Ipilimumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A (JTX-2011) (Experimental): Phase 1 dose escalation and expansion of JTX-2011 by intravenous (IV) infusion
  Interventions: Drug: JTX-2011
- Part B (JTX-2011 + nivolumab) (Experimental): Phase 1 dose escalation and expansion of JTX-2011 by IV infusion in combination with nivolumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Nivolumab
- Part C (JTX-2011) (Experimental): Phase 2 expansion of JTX-2011 by IV infusion
  Interventions: Drug: JTX-2011
- Part D (JTX-2011 + nivolumab) (Experimental): Phase 2 expansion of JTX-2011 by IV infusion in combination with nivolumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Nivolumab
- Part E (JTX-2011 + ipilimumab) (Experimental): Phase 1 dose escalation of JTX-2011 by IV infusion in combination with ipilimumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Ipilimumab
- Part F (JTX-2011 + ipilimumab) (Experimental): Phase 2 expansion of JTX-2011 by IV infusion in combination with ipilimumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Ipilimumab
- Part G (JTX-2011 + pembrolizumab) (Experimental): Phase 1 dose escalation of JTX-2011 by IV infusion in combination with pembrolizumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Pembrolizumab
- Part H (JTX-2011 + pembrolizumab) (Experimental): Phase 2 expansion of JTX-2011 by IV infusion in combination with pembrolizumab by IV infusion
  Interventions: Drug: JTX-2011; Drug: Pembrolizumab

INTERVENTIONS:
Drug: JTX-2011 — Specified dose on specified days
  Other Names: ICOS agonist monoclonal antibody
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part B (JTX-2011 + nivolumab); Part D (JTX-2011 + nivolumab)
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Part E (JTX-2011 + ipilimumab); Part F (JTX-2011 + ipilimumab)
Drug: Pembrolizumab — Specified dose on specified days
  Other Names: Keytruda
  Arms: Part G (JTX-2011 + pembrolizumab); Part H (JTX-2011 + pembrolizumab)

SUMMARY:
JTX-2011-101 is a Phase 1/2, open label, dose escalation and expansion clinical study of JTX-2011 alone and in combination with nivolumab, ipilimumab, or pembrolizumab in adult subjects with advanced and/or refractory solid tumors, to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D), as well as to evaluate preliminary efficacy.

DETAILED DESCRIPTION:
JTX-2011 is an agonist monoclonal antibody that specifically binds to the Inducible CO-Stimulator of T cells (ICOS) to generate an anti-tumor immune response. This is a Phase 1/2, open label, multicenter, dose escalation and expansion, first-in-human (FIH) clinical study to evaluate the safety and tolerability, PK, PD, and preliminary efficacy of the ICOS agonist monoclonal antibody JTX-2011 alone and in combination with nivolumab, ipilimumab, or pembrolizumab in adult subjects with advanced and/or refractory solid tumors. The study will include a dose escalation phase for single agent and the combination therapies, followed by an expansion phase in specified tumor types for single agent and the combination therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing and able to participate and comply with all trial requirements and able to provide signed and dated informed consent prior to initiation of any trial procedures
2. Evaluable or measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, and meet the requirements for the intended study cohort
3. Male or Female ≥ 18 years of age
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1. Subjects with ECOG 2 may be considered for enrollment in Parts C, D, F, and H if approved by Medical Monitor
5. Have a predicted life expectancy of ≥ 3 months
6. Have laboratory values (obtained ≤ 28 days prior to first infusion day) in accordance with the study protocol
7. If medical history of the following, case should be reviewed by the Medical Monitor: prior biliary tract disorders (as based on Hepatobiliary SOC high level terms of: obstructive bile duct disorders, hepatic vascular disorders, structural and other bile duct disorders) or portal hypertension and/or hepatic vascular disorders
8. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to administration of each dose of JTX-2011
9. WOCBP and males with partners of child-bearing potential must agree to use adequate birth control throughout their participation and for 5 months following the last study treatment

Exclusion Criteria:

1. Receiving concurrent anti-cancer treatment (excluding radiation therapy), either approved or investigational
2. Have refused standard therapy
3. Have received anti-cancer therapies listed below within the specified timeframe, or who have ongoing toxicity from prior therapy > Grade 1 according to the Common Terminology for Adverse Events (CTCAE). Exceptions to this are: > Grade 1 toxicities which in the opinion of the Investigator should not exclude the subject (e.g. alopecia, Grade 2 neuropathy, hypo- or hyperthyroidism or other endocrinopathies that are well-controlled with hormone replacement) and are approved by the Medical Monitor.

   1. Have received biologic therapy, including immunotherapy, < 28 days prior to C1D1;
   2. Have received CAR-T therapy;
   3. Have received chemotherapy < 21 days prior to C1D1, or < 42 days for mitomycin or nitrosoureas;
   4. Have received targeted small molecule therapy < 14 days prior to C1D1;
   5. Have undergone organ transplantation including allogeneic or autologous stem-cell transplantation, at any time;
4. Have undergone a major surgery (excluding minor procedures, e.g. placement of vascular access, biopsy, etc.) < 6 months prior to the first day of study treatment, C1D1
5. Have a history of intolerance, hypersensitivity, or treatment discontinuation due to severe immune adverse events on prior immunotherapy, or documented presence of neutralizing anti-drug antibody to nivolumab, ipilimumab, or pembrolizumab. Subjects who discontinued prior immunotherapies for immune-related adverse events that are well-controlled with appropriate treatment may be enrolled if approved by the Medical Monitor.
6. Have a diagnosis of immunodeficiency, either primary or acquired, or treatment with systemic steroids or any other form of immunosuppressive therapy within 7 days prior to C1D1. Exception: inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease as well as a one-time dose of immunosuppressive agents used prophylactically for contrast allergies
7. Have any active disease requiring systemic immunosuppressive treatment
8. Have known severe intolerance to or life-threatening hypersensitivity reactions to humanized monoclonal antibodies or intravenous immunoglobulin preparations; any history of anaphylaxis; prior history of human anti-human antibody response; known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
9. Are symptomatic or have uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation (brain metastases that are stable and asymptomatic, either treated or untreated, will be allowed)
10. Have current second malignancy at other sites, which requires treatment, or in the judgement of the Investigator, may require treatment within the next year. Concurrent malignancies that do not require treatment and are clinically stable are allowed. A past history of other malignancies is allowed as long as the subject is not receiving specific treatment other than hormonal therapy, and, in the judgement of the Investigator, is unlikely to have a recurrence.
11. Have active and clinically relevant bacterial, fungal, or viral infection, including known Hepatitis A, B, or C or human immunodeficiency virus (HIV) (testing not required)
12. Have received live vaccines within past 30 days (inactivated vaccines are allowed; seasonal vaccines should be up to date prior to first infusion day)
13. Women who are pregnant or breastfeeding
14. Have experienced symptomatic cardiac disease that is unresponsive to surgical or medical management
15. Have any medical or social condition that, in the opinion of the Investigator, might place a subject at increased risk, affect compliance, or confound safety or other clinical trial data interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Jounce Therapeutics, Inc.
Locations (16):
- United States (16):
  - Stanford University School of Medicine, Palo Alto, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - The University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute at TriStar Health, Nashville, Tennessee
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment number of 242 is the number of participants who signed the ICF. The number that Started the Participant flow module (218) are those subjects who received any amount of study drug (JTX-2011 and/or nivolumab and/or ipilimumab and/or pembrolizumab). The difference between these two values (24) are the number of patients who screen failed.
Groups:
- Part F (JTX-2011 + Ipilimumab): Phase 2 expansion of JTX-2011 by IV infusion in combination with ipilimumab by IV infusion JTX-2011: Specified dose on specified days Ipilimumab: Specified dose on specified days
- Part H (JTX-2011 + Pembrolizumab): Phase 2 expansion of JTX-2011 by IV infusion in combination with pembrolizumab by IV infusion JTX-2011: Specified dose on specified days Pembrolizumab: Specified dose on specified days
Period: Overall Study
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part F (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab) | Part H (JTX-2011 + Pembrolizumab)
Started | 40 | 31 | 30 | 100 | 11 | 0 | 6 | 0
Completed | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Not Completed | 40 | 29 | 30 | 96 | 11 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Parts F and H were never opened as clinical and translational data from ICONIC suggests that alternative regimens may be preferable to those proposed in Parts F and H.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part F (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab) | Part H (JTX-2011 + Pembrolizumab) | Total
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 0 | 6 | 0 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0
  Between 18 and 65 years | 28 | 27 | 13 | 64 | 7 |  | 2 |  | 141
  >=65 years | 12 | 4 | 17 | 36 | 4 |  | 4 |  | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.94) | 56.2 (9.87) | 64.4 (10.57) | 61.1 (9.65) | 58.8 (9.95) |  | 65.7 (8.77) |  | 60.8 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 13 | 39 | 3 |  | 3 |  | 99
  Male | 18 | 12 | 17 | 61 | 8 |  | 3 |  | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 4 | 0 |  | 0 |  | 14
  Not Hispanic or Latino | 35 | 27 | 26 | 91 | 11 |  | 6 |  | 196
  Unknown or Not Reported | 1 | 0 | 2 | 5 | 0 |  | 0 |  | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0
  Asian | 0 | 2 | 2 | 4 | 0 |  | 0 |  | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 |  | 0 |  | 2
  Black or African American | 6 | 3 | 1 | 5 | 2 |  | 0 |  | 17
  White | 29 | 22 | 22 | 77 | 7 |  | 6 |  | 163
  More than one race | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0
  Unknown or Not Reported | 5 | 4 | 5 | 13 | 1 |  | 0 |  | 28
Region of Enrollment [Number; unit: participants]
  United States | 40 | 31 | 30 | 100 | 11 |  | 6 |  | 218

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with an adverse event occurring from the time of informed consent until resolution or new therapy initiated or for 28 days post final dose if no new therapy is initiated
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 38 | 31 | 30 | 98 | 11 | 6

2. Primary Outcome: Number of Participants With Grade 5 (Fatal) Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with Grade 5 (fatal) treatment emergent adverse events (TEAE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 2 | 2 | 3 | 5 | 0 | 1

3. Primary Outcome: Number of Participants With Grade 4 (Life Threatening) Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with Grade 4 (life threatening) treatment emergent adverse events (TEAE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 1 | 1 | 2 | 4 | 2 | 0

4. Primary Outcome: Number of Participants With Grade 3 (Sever) Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with Grade 3 (severe) treatment emergent adverse events (TEAE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03."
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 17 | 8 | 14 | 43 | 4 | 2

5. Primary Outcome: Number of Participants With Grade 2 (Moderate) Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with Grade 2 (moderate) treatment emergent adverse events (TEAE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 10 | 16 | 8 | 32 | 5 | 3

6. Primary Outcome: Number of Participants With Grade 1 (Mild) Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with Grade 1 (mild) treatment emergent adverse events (TEAE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Time Frame: 46.3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 30 | 100 | 11 | 6
Participants | 8 | 4 | 3 | 14 | 0 | 0

7. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Number of participants with at least one dose limiting toxicity (DLT)
Time Frame: 33 months
Population: Part C and D did not have any participants analyzed for this outcome measure because DLT is only relevant to the Phase 1 parts of study (Part A, Part B, Part E and Part G).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 40 | 31 | 0 | 0 | 11 | 6
Participants | 2 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the proportion of subjects with a Best Overall Response characterized as either a Complete Response (CR) or Partial Response (PR) as defined by RECISTv1.1 guidelines based on investigator's review
Time Frame: 46.5 months
Population: Response Evaluable Set: subjects who received any study drug and have a baseline tumor assessment, and either has at least one post-baseline tumor assessment scan and/or discontinued treatment due to death or disease progression The number of participants analyzed is zero for Part F and Part H because there were no participants enrolled in those two groups of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Participants | 0 | 1 | 1 | 2 | 0 | 0

9. Primary Outcome: Disease Control Rate
Description: Disease Control Rate: Percent Subjects with confirmed Complete Response + confirmed Partial Response + BoR of SD (or unconfirmed complete response or partial response lasting at least 53 days from the date of first dose)
Time Frame: 46.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Participants | 7 | 7 | 3 | 23 | 2 | 4

10. Primary Outcome: Progression Free Survival
Description: Progression free survival, as determined by the Investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Time Frame: 46.5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
months | 2.1 [1.9 to 2.1] | 2.0 [1.8 to 2.2] | 1.9 [1.8 to 2.0] | 2.0 [1.9 to 2.0] | 2.5 [1.3 to 4.1] | 4.0 [1.3 to 10.4]

11. Primary Outcome: 6 Month Landmark Progression Free Survival
Description: Percentage of patients that are progression free at 6 months, estimated by the Kaplan Meier method as the probability of being event-free at 6 months out of the entire 45.5-month primary study period. This method generates survival probability estimates across the Time Frame of the study using all data throughout the course of the trial.
Time Frame: 46.5 months
Population: The 95% CI is not estimable by Kaplan-Meier method for Part E since the probability of event was 0.
Measure: Mean (95% Confidence Interval); unit: Probability of event free at month 6 (%)
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Probability of event free at month 6 (%) | 10.0 [2.1 to 25.3] | 10.2 [2.0 to 26.5] | 4.1 [.3 to 17.6] | 9.1 [3.8 to 17.3] | 0 [NA to NA] — NA Explanation: The 95% CI is not estimable by Kaplan-Meier method since no patients are at risk by the 6 month landmark | 33.3 [1.4 to 75.5]

12. Primary Outcome: 12 Month Landmark Progression Free Survival
Description: Percentage of patients that are progression free at 12 month, estimated by the Kaplan Meier method as the probability of being event-free at 12 months out of the entire 45.5-month primary study period. This method generates survival probability estimates across the Time Frame of the study using all data throughout the course of the trial.
Time Frame: 46.5 months
Measure: Mean (95% Confidence Interval); unit: Probability of event free at month 12(%)
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Probability of event free at month 12(%) | NA [NA to NA] — The 95% CI is not estimable by Kaplan-Meier method since no patients are at risk by the 12 month landmark | 10.2 [2.0 to 26.5] | 4.1 [.3 to 17.5] | 4.6 [1.2 to 11.4] | 0 [NA to NA] — The 95% CI is not estimable by Kaplan-Meier method since no patients are at risk by the 12 month landmark | 0 [NA to NA] — The 95% CI is not estimable by Kaplan-Meier method since no patients are at risk by the 12 month landmark

13. Primary Outcome: Landmark Overall Survival at 6 Months
Description: Percentage of patients that are alive at 6 month, estimated by the Kaplan Meier method as the probability of being event-free at 6 months out of the entire 45.5-month primary study period. This method generates survival probability estimates across the Time Frame of the study using all data throughout the course of the trial.
Time Frame: 46.5 months
Measure: Mean (95% Confidence Interval); unit: Probability of event free at month 6 (%)
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Probability of event free at month 6 (%) | 69.4 [46.8 to 83.9] | 61.8 [40.4 to 77.5] | 47.9 [27.2 to 66.0] | 70.2 [59.1 to 78.8] | 77.8 [36.5 to 93.9] | 66.7 [19.5 to 90.4]

14. Primary Outcome: Landmark Overall Survival at 12 Months
Description: Percentage of patients that are alive at 12 month, estimated by the Kaplan Meier method as the probability of being event-free at 12 months out of the entire 45.5-month primary study period. This method generates survival probability estimates across the Time Frame of the study using all data throughout the course of the trial.
Time Frame: 46.5 months
Measure: Mean (95% Confidence Interval); unit: Probability of event free at month 12(%)
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
Probability of event free at month 12(%) | 12.2 [2.1 to 31.8] | 41.2 [22.2 to 59.3] | 16.0 [4.1 to 34.8] | 40.5 [29.5 to 51.3] | 31.1 [1.5 to 72.3] | 16.7 [.8 to 51.7]

15. Primary Outcome: Overall Survival
Description: The time from first dose date to the date of death for any cause
Time Frame: 46.5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab)
Number analyzed (Participants) | 38 | 29 | 30 | 90 | 9 | 6
months | 7.6 [5.4 to 10.3] | 8.9 [4.7 to 12.7] | 4.9 [3.1 to 9.2] | 9.5 [7.2 to 12.0] | 9.3 [1.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events. | 8.2 [2.9 to NA] — Upper confidence limit is not estimable by Brookmeyer and Crowley method due to insufficient observed events.

ADVERSE EVENTS:
Time Frame: Participants could be monitored for up to 46.5 months (the time from signing consent to 28 days after the last dose is administered)
Description: The first patient signed informed consent on 2016-08-17; 28 days after the last dose was 2020-07-01, therefore AE reporting took place over the course of 46.5 months. AE data was collected via adverse event case report forms using log forms. The number of participants at risk for Serious AEs, All-Cause Mortality, and Other (Not Including Serious) AEs is zero for Part F and Part H because no subjects were enrolled in these parts of the study.
Arm/Group | Part A (JTX-2011) | Part B (JTX-2011 + Nivolumab) | Part C (JTX-2011) | Part D (JTX-2011 + Nivolumab) | Part E (JTX-2011 + Ipilimumab) | Part F (JTX-2011 + Ipilimumab) | Part G (JTX-2011 + Pembrolizumab) | Part H (JTX-2011 + Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 19/40 | 19/31 | 22/30 | 68/100 | 6/11 | 0/0 | 5/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 14/40 | 9/31 | 16/30 | 38/100 | 6/11 | 0/0 | 2/6 | 0/0
Other Adverse Events (participants affected / at risk) | 38/40 | 31/31 | 30/30 | 98/100 | 11/11 | 0/0 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (JTX-2011) (N=40) | Part B (JTX-2011 + Nivolumab) (N=31) | Part C (JTX-2011) (N=30) | Part D (JTX-2011 + Nivolumab) (N=100) | Part E (JTX-2011 + Ipilimumab) (N=11) | Part F (JTX-2011 + Ipilimumab) (N=0) | Part G (JTX-2011 + Pembrolizumab) (N=6) | Part H (JTX-2011 + Pembrolizumab) (N=0)
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Pericarditis
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 5 | 0 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | NA | 1 | NA
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | NA | 0 | NA
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | NA | 0 | NA
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | 0 | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1 | NA | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | NA | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | NA | 0 | NA
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | NA | 0 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | NA | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | NA | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | NA | 0 | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 0 | NA | 0 | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0 | NA | 0 | NA
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | NA | 0 | NA
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 0 | NA | 0 | NA
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | NA | 0 | NA
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | NA | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Hypercalcaemia (General disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | NA | 1 | NA
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3 | 0 | NA | 0 | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | NA | 0 | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | NA | 0 | NA
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | NA | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | 0 | NA
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | NA | 0 | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | NA | 1 | NA
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | NA | 0 | NA
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | NA | 0 | NA
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | NA | 0 | NA
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | NA | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (JTX-2011) (N=40) | Part B (JTX-2011 + Nivolumab) (N=31) | Part C (JTX-2011) (N=30) | Part D (JTX-2011 + Nivolumab) (N=100) | Part E (JTX-2011 + Ipilimumab) (N=11) | Part F (JTX-2011 + Ipilimumab) (N=0) | Part G (JTX-2011 + Pembrolizumab) (N=6) | Part H (JTX-2011 + Pembrolizumab) (N=0)
Nausea (Gastrointestinal disorders) | 10 | 14 | 8 | 32 | 2 | 0 | 2 | 0 — Intermittent nausea
Vomiting (Gastrointestinal disorders) | 4 | 8 | 7 | 16 | 2 | NA | 2 | NA
Diarrhea (Gastrointestinal disorders) | 7 | 4 | 5 | 18 | 3 | NA | 1 | NA
Constipation (Gastrointestinal disorders) | 3 | 8 | 6 | 14 | 4 | NA | 2 | NA
Abdominal pain (Gastrointestinal disorders) | 8 | 2 | 8 | 8 | 2 | NA | 1 | NA
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 2 | 12 | 1 | NA | 1 | NA
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 3 | 4 | 0 | NA | 0 | NA
Ascites (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0 | NA | 0 | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 0 | NA | 0 | NA
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 0 | NA | 0 | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | NA | 0 | NA
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | NA | 2 | NA
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | NA | 0 | NA
Retching (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | NA | 0 | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | NA | 0 | NA
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Fatigue (General disorders) | 9 | 10 | 15 | 37 | 7 | NA | 2 | NA
Pyrexia (General disorders) | 6 | 5 | 4 | 24 | 0 | NA | 2 | NA
Chills (General disorders) | 6 | 3 | 1 | 13 | 2 | NA | 2 | NA
Oedema peripheral (General disorders) | 2 | 3 | 6 | 5 | 1 | NA | 0 | NA
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 5 | 1 | NA | 1 | NA
Chest discomfort (General disorders) | 0 | 2 | 0 | 2 | 0 | NA | 0 | NA
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 1 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 8 | 5 | 10 | 29 | 6 | NA | 3 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 5 | 17 | 2 | NA | 3 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 4 | 2 | 8 | 2 | NA | 1 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 8 | 3 | NA | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 6 | 6 | 1 | NA | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 7 | 1 | NA | 1 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 5 | 0 | NA | 1 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 9 | 1 | NA | 0 | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 2 | NA | 0 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1 | NA | 0 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1 | NA | 0 | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | NA | 1 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 6 | 23 | 2 | NA | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 22 | 2 | NA | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 5 | 1 | NA | 1 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 0 | NA | 0 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 1 | 0 | NA | 0 | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 0 | NA | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 0 | NA | 0 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | NA | 0 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | NA | 0 | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | NA | 1 | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 18 | 2 | NA | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 13 | 2 | NA | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 10 | 0 | NA | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 8 | 1 | NA | 0 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 4 | 0 | NA | 0 | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 6 | 0 | NA | 0 | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 0 | NA | 1 | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 0 | NA | 0 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | NA | 1 | NA
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 4 | 12 | 2 | NA | 0 | NA
Weight decreased (Investigations) | 1 | 0 | 5 | 14 | 2 | NA | 1 | NA
Alanine aminotransferase increased (Investigations) | 5 | 2 | 4 | 4 | 0 | NA | 0 | NA
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 3 | 6 | 1 | NA | 0 | NA
Blood bilirubin increased (Investigations) | 2 | 1 | 2 | 5 | 0 | NA | 1 | NA
Blood creatinine increased (Investigations) | 1 | 3 | 1 | 1 | 1 | NA | 0 | NA
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 2 | 2 | NA | 0 | NA
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 3 | 0 | NA | 1 | NA
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | 1 | NA
Electrocardiogram QT prolonged (Investigations) | 3 | 0 | 0 | 0 | 0 | NA | 0 | NA
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | 0 | NA
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
Dizziness (Nervous system disorders) | 4 | 0 | 8 | 13 | 0 | NA | 1 | NA
Headache (Nervous system disorders) | 4 | 2 | 1 | 13 | 2 | NA | 2 | NA
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 0 | 3 | 0 | NA | 1 | NA
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | NA | 0 | NA
Balance disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | NA | 1 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | NA | 1 | NA
Urinary tract infection (Infections and infestations) | 1 | 3 | 2 | 9 | 1 | NA | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 2 | 3 | 0 | NA | 0 | NA
Oral candidiasis (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | NA | 0 | NA
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | NA | 0 | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | NA | 1 | NA
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 9 | 0 | NA | 2 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 6 | 0 | NA | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 6 | 0 | NA | 0 | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | NA | 1 | NA
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | NA | 0 | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | NA | 0 | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | 0 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 9 | 3 | 16 | 2 | NA | 2 | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | 0 | NA
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Anaemia (Blood and lymphatic system disorders) | 9 | 4 | 7 | 11 | 3 | NA | 4 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | NA | 0 | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Insomnia (Psychiatric disorders) | 3 | 1 | 1 | 11 | 0 | NA | 0 | NA
Anxiety (Psychiatric disorders) | 2 | 2 | 1 | 5 | 0 | NA | 2 | NA
Confusional state (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | NA | 0 | NA
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | NA | 1 | NA
Hypertension (Vascular disorders) | 3 | 1 | 2 | 7 | 0 | NA | 0 | NA
Hypotension (Vascular disorders) | 2 | 1 | 1 | 5 | 0 | NA | 2 | NA
Hot flush (Vascular disorders) | 1 | 0 | 0 | 4 | 1 | NA | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 0 | NA | 0 | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | NA | 1 | NA
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | NA | 0 | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | NA | 1 | NA
Tachycardia (Cardiac disorders) | 3 | 2 | 2 | 5 | 0 | NA | 0 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 4 | 0 | NA | 0 | NA
Hyerthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | NA | 0 | NA
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | NA | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication ("pub.") can be restricted until the 1st to occur of (a) pub. of the clinical trial results, or (b) 18 mo's after the Primary Completion Date. Pub. rights depend on PI conducting the study in compliance with the Protocol, that the pub. is made in a recognized journal or conference, and makes use of all study data. The Sponsor can require removal of Sponsor's confidential information from any pub. and can defer pub. for up to an add'l 60 days to file a related patent application.

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT02904226/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT02904226/SAP_001.pdf